CLINICAL TRIAL: NCT06940765
Title: Adipose-Derived Stromal Vascular Fraction Cell Therapy to Treat Post COVID-19 Respiratory Distress - An Early Feasibility Study
Brief Title: Autologous Adipose-derived Stromal Vascular Fraction for Treatment of Post COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No study sites established
Sponsor: GID BIO, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIDC19-2
Record Dates: First submitted 2021-08-19; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open Label Treatment Arm (Experimental): A single intravenous injection of autologous adipose-derived SVF for treatment of continuing respiratory distress after recovery from COVID-19 for reintroduction to the same patient during a single surgical procedure.
  Interventions: Device: GID SVF-2 Device System

INTERVENTIONS:
Device: GID SVF-2 Device System — The GID SVF-2 device is indicated for use for harvesting, filtering, separating, and concentrating autologous stromal vascular fraction cells from adipose tissue.

SUMMARY:
This study is an early feasibility study to evaluate the safety of a single intravenous injection of autologous adipose-derived SVF produced using the GID SVF-2 device system for treatment of continuing respiratory distress after recovery from COVID-19.

DETAILED DESCRIPTION:
The GID SVF-2 device is indicated for use for harvesting, filtering, separating, and concentrating autologous stromal vascular fraction cells from adipose tissue for reintroduction to the same patient during a single surgical procedure for treatment of continuing respiratory distress after recovery from COVID-19.

The primary objective of this study is to evaluate the safety of a single intravenous injection of autologous adipose-derived SVF for treatment of continuing respiratory distress after recovery from initial COVID-19 infection.

The secondary objective is preliminary assessment of feasibility of a single intravenous injection of autologous adipose-derived SVF for treatment of continuing respiratory distress after recovery from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects that are ambulatory and previously hospitalized for a confirmed diagnosis of COVID-19 using RT-PCR test
2. Male or female subjects between the ages of 18-75
3. SpO2 > 92% on room air
4. Subjects with BMI ≥22
5. Subjects with Forced Vital Capacity (FVC) ≥ 40% predicted and ≤ 70% predicted
6. Subjects with DLCO ≥ 20% predicted and ≤ 70% predicted
7. Study Subjects must be willing to voluntarily give written Informed Consent to participate in the study before any study procedures are performed
8. Subjects with the ability to speak, read and understand English
9. Subjects with the ability to complete follow up as specified in the protocol

Exclusion Criteria:

1. Subjects taking immunosuppressive drugs
2. Subjects with history of lung malignancy
3. Subjects allergic to lidocaine or epinephrine
4. Women that are pregnant or planning to become pregnant during the study
5. Women that are lactating
6. Women on hormonal contraceptives in the past 30 days
7. Women currently on hormone replacement therapy
8. Subjects with chronic kidney disease Stage 4 and Stage 5
9. Subjects with a history of pulmonary embolism
10. Subjects with a history of anti-phospholipid syndrome
11. Subjects participating in any other clinical study
12. Subjects with history of deep vein thrombosis
13. Subjects with history of Cirrhosis with Pugh classification of B or C
14. Subjects on hemodialysis
15. Subjects with organ dysfunction or predisposed to organ dysfunction (i.e., pre-dialysis & orthopnea)
16. Subjects with a history of prior clotting disorders or thrombotic syndrome
17. Subjects with myocardial infarction within the past 2 months
18. Subjects with blood pressure <85/50 mmHg or >160/100 mmHg or mean arterial pressure <60 mmHg or >120 mmHg
19. Subjects with a history of drug or alcohol abuse
20. Pulse <50 bpm or >140 bpm
21. Cardiac rhythm showing rapid atrial fibrillation with heart rate >120 bpm or ventricular tachycardia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Safety- adverse events | Baseline to 3 months post treatment
  Evaluation of type and frequency of adverse events.

SECONDARY OUTCOMES:
Pulmonary Function - SpO2(%) | Baseline to 3 months post treatment
  Changes in the following test:
  SpO2 level (%): Oxygen saturation Percent of hemoglobin binding sites in arterial blood occupied by oxygen (%sat)
Pulmonary Function - Forced Vital Capacity | Baseline to 3 months post treatment
  Changes in the following test:
  Pulmonary Function (Forced Vital Capacity): Lung volume in liters and percent of predicted
Pulmonary Function - Carbon Monoxide diffusing Capacity | Baseline to 3 months post treatment
  Changes in the following tests:
  Carbon Monoxide diffusing Capacity (DLCO): ml/min/mm Hg and percent of predicted

CONTACTS AND LOCATIONS:
Overall Officials: William Cimino, Phd, Study Chair — GID BIO

IPD SHARING:
Plan to Share IPD: No